CLINICAL TRIAL: NCT00818272
Title: Remicade Safety Line (Crohn's Disease)
Brief Title: Remicade Safety Line (Crohn's Disease)(Study P03288)(COMPLETED)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: P03288
Record Dates: First submitted 2009-01-06; First posted 2009-01-07 (Estimated); Results first posted 2012-02-01 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-09

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Remicade (infliximab): Participants with confirmed diagnosis of active Crohn's disease.
  Interventions: Biological: Remicade (infliximab)

INTERVENTIONS:
Biological: Remicade (infliximab) — Participants with confirmed diagnosis of severe active Crohn's disease (CD) and participants suffering from fistulae who do not respond sufficiently to a complete and adequate therapy with a conventional treatment received infliximab administration as intravenous (IV) infusion over a period of two hours. Dosage and infusion intervals were employed in accordance to the Summary of Product Characteristics (SmPC): 5 mg/kg body weight at week 0 of infliximab therapy with additional infusions of 5 mg/kg at week 2 and week 6 after the initial dose, followed by infusions every 8 weeks (maintenance) or if signs and symptoms of the disease recur (readministration).
  Other Names: Remicade; SCH 215596

SUMMARY:
This observational study is in line with the German educational plan with the aim to implement a tool to increase and monitor the awareness for tuberculosis screening and to reinforce the patient eligibility for a treatment with Remicade according to the Summary of Product Characteristics (SmPc).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Crohn's disease.

Exclusion Criteria:

* As per SmPC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with Crohn's disease.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2002-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Infliximab: Participants with confirmed diagnosis of severe active Crohn's disease (CD) and participants suffering from fistulae who do not respond sufficiently to a complete and adequate therapy with a conventional treatment received infliximab administration as intravenous (IV) infusion over a period of two hours. Dosage and infusion intervals were employed in accordance to the Summary of Product Characteristics (SmPC): 5 mg/kg body weight at week 0 with additional infusions of 5 mg/kg at week 2 and week 6 after the initial dose, followed by infusions every 8 weeks (maintenance) or if signs and symptoms of the disease recur (readministration).
Period: Overall Study
Arm/Group | Infliximab
Started | 148
Completed | 74
Not Completed | 74

BASELINE CHARACTERISTICS:
Groups:
- Infliximab: Participants with confirmed diagnosis of severe active CD and participants suffering from fistulae who do not respond sufficiently to a complete and adequate therapy with a conventional treatment received infliximab administration as IV infusion over a period of two hours. Dosage and infusion intervals were employed in accordance to the SmPC: 5 mg/kg body weight at week 0 with additional infusions of 5 mg/kg at week 2 and week 6 after the initial dose, followed by infusions every 8 weeks (maintenance) or if signs and symptoms of the disease recur (readministration).
Arm/Group | Infliximab
Number analyzed (Participants) | 148
Age, Continuous [Mean (Standard Deviation); unit: years] — Age data collected for 147 participants
  years | 36.01 (11.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84
  Male | 64

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had the Mendel Mantoux Test as the First Screening Test for Active or Latent Tuberculosis (TB) Before Starting Treatment
Description: In order to increase the attending physician's awareness of the required tuberculosis screening and to support the screening itself, tuberculosis screening was performed and documented before treatment administration (baseline). The number of participants who had the Mendel Mantoux test (tuberculin sensitivity skin test by intradermal injection) as the first screening test was presented in three categories:
  * Yes
  * No
  * Missing (represents no entry, but may mean another test was performed as first screening test and documented)
Time Frame: Baseline
Measure: Number; unit: Participants
Arm/Group | Infliximab
Number analyzed (Participants) | 148
Participants
  Yes | 92
  No | 53
  Missing | 3

2. Secondary Outcome: Assessment of Disease Activity by Means of the Crohn's Disease Activity Index (CDAI) at the Time of Enrollment and at the First Infusion
Description: The CDAI score is used to quantify the symptoms of participants with CD. The CDAI incorporates 8 items added together that are indicators of disease severity. Scores range from 0 to 600; higher scores indicate worse disease activity. Participants with scores below 150 have inactive disease whereas those with scores above 450 are considered critically ill. A decrease in CDAI over time indicates improvement in disease activity. CDAI was calculated at the time of enrollment (baseline) and at the time of first infusion.
Time Frame: Baseline and time of first Infusion
Population: Data was analyzed for all CD participants whose data had been entered in the database and finalized by signature of the physician. 90 out of 148 participants available at enrollment completed the CDAI and 42 out of the 128 available participants at first infusion after screening (beginning of 2 year observation period) completed the CDAI.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Infliximab
Number analyzed (Participants) | 148
Score on a scale
  CDAI at Time of Enrollment (N=90) | 302.67 (126.22)
  CDAI at First Infusion (N=42) | 323.21 (131.45)

3. Primary Outcome: Number of Participants Who Had the Tine Test as the First Screening Test for Active or Latent Tuberculosis Before Starting Treatment
Description: In order to increase the attending physician's awareness of the required tuberculosis screening and to support the screening itself, tuberculosis screening was performed and documented before treatment administration (baseline). The number of participants who had the Tine test (multiple puncture tuberculin skin test) as the first screening test was presented in three categories:
  * Yes
  * No
  * Missing (represents no entry, but may mean another test was performed as first screening test and documented)
Time Frame: Baseline
Measure: Number; unit: Participants
Arm/Group | Infliximab
Number analyzed (Participants) | 148
Participants
  Yes | 40
  No | 105
  Missing | 3

4. Primary Outcome: Number of Participants Who Had the In-vitro TB Test as the First Screening Test for Active or Latent Tuberculosis Before Starting Treatment
Description: In order to increase the attending physician's awareness of the required tuberculosis screening and to support the screening itself, tuberculosis screening was performed and documented before treatment administration (baseline). The number of participants who had the in-vitro TB test (cellular blood test, i.e. gamma interferon release assays) as the first screening test was presented in three categories:
  * Yes
  * No
  * Missing (represents no entry, but may mean another test was performed as first screening test and documented)
Time Frame: Baseline
Measure: Number; unit: Participants
Arm/Group | Infliximab
Number analyzed (Participants) | 148
Participants
  Yes | 0
  No | 90
  Missing | 58

5. Primary Outcome: Number of Participants Who Had a Chest X-ray as Part of TB Screening for Active or Latent Tuberculosis Before Starting Treatment
Description: In order to increase the attending physician's awareness of the required tuberculosis screening and to support the screening itself, tuberculosis screening was performed and documented before treatment administration (baseline). If done according to guidelines, complete TB screening comprised a TB screeing test and a chest X-ray. The number of participants who had a frontal chest X-ray was presented in three categories:
  * Yes
  * No
  * Missing
Time Frame: Baseline
Measure: Number; unit: Participants
Arm/Group | Infliximab
Number analyzed (Participants) | 148
Participants
  Yes | 131
  No | 14
  Missing | 3

ADVERSE EVENTS:
Arm/Group | Infliximab
Serious Adverse Events (participants affected / at risk) | 0/148
Other Adverse Events (participants affected / at risk) | 0/148

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Trial results belong to the SPONSOR only, all investigators are not allowed to publish trial results without permission of the SPONSOR.